CLINICAL TRIAL: NCT04404270
Title: Study of SARS-CoV2 Virus (COVID-19) Seroprevalence in the Population of Creil Air Force Base (BA110)
Acronym: EpiCovCreil
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-22; 2020-A01368-31 (Other: IDRCB)
Record Dates: First submitted 2020-05-25; First posted 2020-05-27 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Sars-CoV2
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Anti-SARS-CoV2 Serology — The anti-SARS-CoV2 serological status will be measured on a blood sample collected at Day 0.
Behavioral: Questionnaire — Epidemiological data will be collected in a questionnaire that will be filled by participants at Day 0 (Visit 1), after 3 months (Visit 2) and after 9 months (Visit 3).
  The questionnaire includes:
  * medical data (height, weight, smoking, history of intense stress);
  * socio-demographic data (age, gender, civil/military status, function/occupation, rank category, army, family status/home composition, housing conditions, etc.);
  * clinical data : history of symptoms suggestive of COVID-19 in the last 3 months, current symptoms suggestive of COVID-19;
  * use of care, hospitalization, work stoppage in the last 3 months;
  * contact with people who are symptomatic or proven COVID-19.
Diagnostic Test: Anti-SARS-CoV2 serological controls and serum neutralization — Serological controls and a serum neutralization test will be performed on blood samples collected 3 months (Visit 2) and 9 months (Visit 3) after Day 0, respectively.

SUMMARY:
In mid-February 2020, within the Oise (France) cluster, a case of COVID-19 disease caused by a SARS-CoV2 infection was described among the personnel of the Creail Air Force Base (BA110). This resulted in the beginning of an epidemic controlled by epidemiological measures. One month later, containment measures were taken at the national level, measures that also applied to BA110 personnel. These personnel, exposed to both the initial phase of the epidemic and national protection measures, represent an extremely interesting population for understanding the epidemiological dynamics of the virus, particularly at a time when France is lifting the containment measures. It becomes extremely important to understand the levers of viral spread in order to adjust the health measures to be maintained as best as possible.

The main objective of this study is to determine the extent of virus diffusion in this highly circulating population, as evidenced by several identified cases of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Active military or civilian defence personnel working on the Creil Air Force Base (BA110) during the period of interest (from February 1st 2020 to the end of the study)

Exclusion Criteria:

* Contraindication to blood sampling
* Pregnant, parturient, breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The eligible population is composed of all civilian and military personnel working on the Creil Air Force Base (BA110) or having worked on BA110 as a permanent personnel since February 1st 2020, including the people working in satellite units such as the "Groupement de soutien de base de Défense" de Creil ("Creil Defence Base Support Group") or the 3/60 Esterel squadron.
Sampling Method: Non-Probability Sample
Enrollment: 1146 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Proportion anti-SARS-CoV2 seropositive | Day 0
  The percentage of the study population with positive serological status will be determined. ELISA serology test will be used to detect anti-SARS-CoV2 antibodies (IgG and IgM) at Day 0

SECONDARY OUTCOMES:
Proportion of asymptomatic anti-SARS-CoV2 seropositive participants | Day 0
  Among anti-SARS-CoV2 seropositive participants, the percentage of asymptomatic participants will be determined. COVID-19 symptoms will be measured using a questionnaire.
Agreement between the anti-SARS-CoV2 serological results obtained using two different techniques (detecting the presence of different antibodies) | Day 0
  The serological results obtained using the reference ELISA test results (detecting the presence of IgG and IgM antobodies) and using a second ELISA test detecting the presence of antibodies specifically directed against the Receptor Binding Domain and the Spike protein trimer of SARS-CoV2 virus will be compared.
Proportion of serum neutralization positive | Day 0
  Among anti-SARS-CoV2 seropositive participants, the percentage of participants with a positive response to serum neutralization will be determined.
Change of antibody level over time | 3 months and 9 months after Day 0
  The evolution of the antibody level over time will be determined using repeated serodiagnoses at 3 and 9 months.

CONTACTS AND LOCATIONS:
Locations (1):
- 24e antenne médicale de Creil, Creil, France